CLINICAL TRIAL: NCT06813053
Title: A Novel Decision Aid for Early Stage Breast Cancer Patients Choosing Between Lumpectomy and Mastectomy: a Pilot Study
Brief Title: A Novel Patient Decision Aid for Surgical Treatment Options in Early-Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Association of Academic Surgery (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-0577.cc; NCT-2025-02972 (Other: CTRP)
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Early-Stage; Newly Diagnosed
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Newly detected, early stage breast cancer patients in the treatment group will be provided an electronic copy of the DA for their reference via email.
  Interventions: Other: Decision Aid (DA)
- Control Group (Placebo Comparator): Newly diagnosed, early stage breast cancer patients in the control group will be provided an electronic copy of an alternative educational pamphlet discussing surgical options for breast cancer.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Other: Decision Aid (DA) — Tools designed to foster shared decision-making by contextualizing the risks and benefits of treatment options around the patient's personal values, thereby allowing them to weigh personal preferences when making treatment decisions. The study team has developed a prototype DA incorporating longitudinal institutional QoL data among patients who have undergone breast cancer surgery .
  Arms: Interventional Group
Other: Standard of Care (SOC) — Electronic copy of an alternative educational pamphlet discussing surgical options for breast cancer.
  Arms: Control Group

SUMMARY:
This is a study to assess the feasibility and acceptability of a novel decision aid (DA) in a newly diagnosed, early-stage breast cancer population. Insights gained from patient feedback and the implementation process will be used to improve the information delivered in the decision aid itself and to plan for a larger scale trial to compare the decision aid to standard of care.

DETAILED DESCRIPTION:
This pilot study will utilize several tools and instruments to measure various aspects of of the implementation of the decision aid. 1. BREAST-Q patient-Reported Outcomes, 2. Ottawa Decision Aid Evaluation Measures, 3. Health Literacy Assessments, 4. Distress Screening Tools, 5. Web-Based Surveys, 6. Semi-Structured Interviews.

ELIGIBILITY:
Inclusion Criteria:

* Adult women age 18-100
* English speaking
* Clinical stage 0-III breast cancer
* Eligible for both lumpectomy and mastectomy

Exclusion Criteria:

* Prior surgical consultation regarding treatment options for breast cancer
* Previous history of breast cancer
* Requires neoadjuvant chemotherapy prior to surgical intervention

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of prospectively providing a novel DA to early stage breast cancer patients | 1 year
  Monitor the recruitment process of eligible patients. Including tracking how many patients are approached, how many participate and how effective the decision aid engages patient in the decision making process. High participation and engagement indicates a successful implementation. Compare clinician reported length of encounter between interventions as a balancing measure.
Evaluate how well patients receive the decision aid | 1 year
  Use the validated and accepted Ottawa Decision Aid metrics to assess decision quality, decisional conflict, acceptability, and regret. Conduct semi-structured interviews to gather additional qualitative data regarding the patient experience, and use feedback to modify and improve the content and design of the Decision Aid.

SECONDARY OUTCOMES:
Maximize patient engagement with the decision aid | 1 year
  Optimal timing and mode of delivery will be determined by the engagement of patients with the decision aid (DA) based on the time the DA was offered. Qualitative feedback from semi-structured interviews will provide additional context for engagement with paper versus digital copies, and engagement prior to versus after meeting with the surgeon.
Obtain pilot data for a large scale randomized controlled trial comparing use of the decision aid to standard of care in early-stage breast cancer patients. | 1 year
  Patient-reported Decision Aid Acceptability, Decision Quality, Self Efficacy, Decision Conflict, and Decision Regret (from the Ottawa Decision Aid Measures) as well as Patient-reported distress will be compared between intervention groups. Differences in these key outcomes will be used to perform a power analysis to determine optimal enrollment size for a large scale multicenter randomized controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Tevis, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - Universtiy of Colorado Hospital, Aurora, Colorado
  - UCHealth Cherry Creek Medical Center, Denver, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado